CLINICAL TRIAL: NCT06981988
Title: A Study to Explore the Dosage and Efficacy of Linperlisib in Combination With Rituximab and to Validate the Efficacy of Linperlisib in Patients With Relapsed/Refractory Indolent NHL
Brief Title: A Study of Linperlisib (YY-20394) in Combination With Rituximab in Patients With Relapsed/Refractory Indolent NHL
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS3536-III-301
Record Dates: First submitted 2023-04-04; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Relapsed/Refractory Indolent NHL
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Linperlisib + Rituximab (Experimental)
  Interventions: Drug: Linperlisib ； Rituximab

INTERVENTIONS:
Drug: Linperlisib ； Rituximab — Linperlisib ； Rituximab

SUMMARY:
The study is being conducted to evaluate the reasonable dosage, efficacy and safety of Linperlisib in combination with rituximab in subjects with relapsed/refractory (R/R) indolent non-hodgkin lymphoma(NHL) in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Patients received at least 1 lines of systemic therapy
2. Previously received anti- CD20 treatment
3. Subjects must have at least one bi-dimensionally measurable lesion (nodal site Ldi > 1.5 cm or extranodal site Ldi > 1.0cm)
4. Patients must have an acceptable organ function

Exclusion Criteria:

1. Previously treated with PI3K inhibitors
2. Unresolved toxicity of CTCAE grade > 1 from prior anti-lymphoma therapy
3. Chemotherapy or other antitumor therapy within 14 days before starting cycle one
4. Significant concurrent medical disease or condition which according to the investigators' judgement
5. Active hepatitis B, C or HIV infection
6. Infection requiring treatment 2 weeks prior to the first dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
MTD （Maximum tolerated dose）of Linperlisib（Stage 1） | Subjects are evaluated for DLTs during the first 28-day cycle
RP2/3D（Recommended Phase II/III Dose) of Linperlisib （Stage 1） | The RP2/3D for Phase 2/3 will be selected at the end of Phase 1b, approximately 2 years
Complete response rate (CRR) assessed by Investigator（Stage 2） | up to 5 years
Progression-free Survival assessed by Investigator （Stage 2） | up to 5 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) assessed by Investigator | up to 5 years
Duration of response (DOR) assessed by Investigator | up to 5 years
Incidence of Adverse Events (Linperlisib when combined with Rituximab) | up to 5 years

IPD SHARING:
Plan to Share IPD: Undecided